CLINICAL TRIAL: NCT07014696
Title: Investigation of the Effects of PNF and Kinesiological Taping on Hand Function in Hemiplegic Stroke Patients Based on the ICF Framework
Brief Title: ICF-Based Effects of PNF and Kinesio Taping on Hand Function in Hemiplegic Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Collaborators: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Elif Önder, Physical therapist, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2024000565-1
Record Dates: First submitted 2025-05-20; First posted 2025-06-11 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Hemiplegia; Hemiplegia Due to Stroke; Hand Functionality; Upper Extremity; Proprioceptive Neuromuscular Facilitation; Kinesio Taping
Keywords: hand functionality; hemiplegia; hemiplegia due to stroke; upper extremity; ICF; Proprioceptive neuromuscular facilitation; kinesio taping
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Intervention Model Description: Treatment Method: Patients who continue the rehabilitation program due to hemiplegic stroke and meet the inclusion criteria will be treated. The treatment will be applied in addition to the conventional physiotherapy program for 24 sessions, 3 days a week for 8 weeks.
  Group 1: PNF application Group (n: 18): Conventional Physiotherapy + PNF application Group 2: KB application Group (n: 18): Conventional Physiotherapy + KB application Group 3: PNF+KB application Group (n: 18): Conventional Physiotherapy + PNF + KB application
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: PNF application Group (Experimental): In the PNF method to be applied to the first group, the subjects will be in a sitting position. The application will be made to the fingers, wrist and forearm in both D1 and D2 direction flexion and extension patterns. The techniques will start by using rhythmic initiation, then the combination of isotonics, dynamic-opposite, rhythmic stabilization and muscle-relaxation will be determined. The movements will be done with 10 repetitions and rest in between. The exercises will continue for 8 weeks, 3 days a week.After all applications, conventional treatment will be applied to all three groups.
  Interventions: Procedure: PNF application Group
- Group 2: KB Application Group (Experimental): In the taping treatment to be applied to the second group, taping will be applied starting from the fingers to the elbow with kinesiology taping. Taping will be done 3 days a week and the tape will remain on the patient for 2 days. Exercises will continue 3 days a week for 8 weeks. After all applications, conventional treatment will be applied to all three groups.
  Interventions: Procedure: KB application Group
- Group 3: PNF+KB application Group (Experimental): The third group will be applied both PNF and taping. Exercises will continue 3 days a week for 8 weeks. After all applications, conventional treatment will be applied to all three groups.
  Interventions: Procedure: PNF+KB application Group

INTERVENTIONS:
Procedure: PNF application Group — PNF Application; in the application method, the subjects will be in a sitting position. The application will be made to the fingers, wrist and forearm in both D1 and D2 directions in flexion and extension patterns. The techniques will start using rhythmic initiation, then the combination of isotonics, dynamic-opposite, rhythmic stabilization and muscle-relaxation are determined. The movements will be made in 10 repetitions with rest in between (Saklecha et al., 2023).
  Arms: Group 1: PNF application Group
Procedure: KB application Group — KB Application; In the taping treatment to be applied, taping will be applied starting from the fingers and up to the elbow with kinesiology taping (Huang et al., 2019). Taping will be done 3 days a week and the tape will remain on the patient for 2 days.
  Arms: Group 2: KB Application Group
Procedure: PNF+KB application Group — PNF+ KB Application; In this application, both PNF and taping will be applied. After each application, conventional treatment will be applied to all three groups at the end of each session. When all treatments are completed, re-evaluations will be made by the blind physiotherapist
  Arms: Group 3: PNF+KB application Group

SUMMARY:
This clinical trial aims to compare the effects of kinesio taping and PNF on hemiplegic hand functions. In addition, the effects of these applications on body structure, activity, and participation will be examined. The main questions it aims to answer are:

Do kinesio taping and PNF applications have different effects on hemiplegic hand function? Are kinesio taping and PNF applications effective in body structure, activity, and participation? The researchers will compare the advantages of kinesio taping and PNF applications over each other.

Participants:

Kinesio taping and/or PNF applications will be applied 3 days a week for 8 weeks.

Tests will be performed on the first and last day of the study to evaluate hand functions.

DETAILED DESCRIPTION:
This study aims to investigate the effects of proprioceptive neuromuscular facilitation and kinesiology taping on hand functions in hemiplegic stroke patients. In order to evaluate functionality, it will be evaluated with the Box block test, Fugl Meyer upper extremity test, ARAT, and nine-hole peg test. In order to examine the cases within the scope of functionality, disability, and health international classification (ICF), environmental quality scale, upper extremity motor activity diary-28, stroke impact scale, and social adaptation scale will be evaluated.

Stroke is the second leading cause of death and disability among adults over the age of 60 worldwide. Approximately 17 million people have a stroke every year in the world and 140 thousand people in our country. Data from all over the world also reveal that the incidence of stroke will increase in the coming years. By definition, stroke is a clinical condition that develops after focal infarction or hemorrhage in the cerebral cortex, cerebellum and spinal cord, causes focal neurological dysfunction, can last 24 hours or longer and can even result in death. After a stroke, the surrounding brain tissue is deprived of oxygen and essential nutrients, and if left untreated, it can lead to permanent tissue damage, including neuronal cell death. Damages that occur after a stroke cause motor, sensory, and cognitive impairments in individuals; upper extremity dysfunction, balance, and walking difficulties, causing people to be dependent on various degrees in their daily life activities. Post-stroke disability reduces the quality of life of the individual and their relatives, affecting their lives. It also causes both socioeconomic and social problems. Approximately 50-75% of those affected in the early post-stroke period experience upper extremity impairment, and a large portion of them will live with long-term upper extremity impairment. Although most individuals regain walking function after stroke, very few individuals are able to use their upper extremities, especially their hands, at a fully functional level. Upper extremity function after stroke is among the main causes of long-term disability. This is because the natural recovery of upper extremity function is generally more limited than that of the lower extremity. Impaired use of the upper extremity persists in approximately 60% of patients even 6 months after stroke. Exercise interventions are necessary to improve upper extremity motor functions and activities of daily living (ADL) in stroke patients, because persistent upper extremity dysfunction is strongly associated with decreased activities of daily living and poor quality of life after stroke.

Abnormal synergies occur in the extremities of patients who have had a stroke. The literature has described two main synergies for the upper extremity: Flexion or extension synergy patterns. These synergies in the upper extremity and hand lead to loss of mobility, interfere with activities of daily living including dressing and hygiene, may cause skin breakdown, and may cause pain. Over time, weakness in the hemiparetic hand, motor disorders caused by abnormal synergies, and permanent spasticity begin to cause secondary changes in the musculoskeletal system that may limit the use of the arm and hand and affect functional mobility; soft tissue shortening and contracture formation may be observed. There is a wide range of treatments for upper extremity recovery following stroke. In these methods, integrated treatments are recommended for both the hand and arm. Upper limb rehabilitation aims to provide all possible means to regain lost function and increase the autonomy of stroke patients, taking into account any remaining impairments and disabilities. Carr and Shepherd suggested that poor recovery in the upper limb may result from the direct effects of stroke as well as from inadequate, inappropriate or incorrect therapeutic interventions. However, little information is available to explain what best represents the "optimal treatment". The chosen treatment modality may be directed at a specific impairment (e.g. muscle weakness) or functional movements (e.g. grasping and letting go activity). These treatment modalities may be used separately or combined to address the multifactorial impairments that may arise following stroke, i.e. primary problems and secondary complications. Therefore, it should be noted that upper extremity rehabilitation after stroke will involve a complex intervention that requires the cooperation of the patient, caregivers, and the rehabilitation team.

Neuromuscular therapies, one of the approaches used in the treatment of stroke, include multiple methods. In recent years, activities related to the recovery of motor functions have become the focus of research by scientists dedicated to the development of the topic of brain plasticity, which allows a person to adapt to the environment through learning and self-repair after damage. A typical example of neural plasticity is the recovery process after ischemic stroke, which initiates the reorganization of the central nervous system and the assumption of some functions by undamaged parts of brain structures. Reorganization also involves the expansion of cortical areas that provide the neural substrate for the recovery or adaptation of motor activities after damage. The results of studies on brain plasticity have revealed that the proprioceptive neuromuscular facilitation (PNF) technique, one of the neuromuscular treatments, provides the development of neurorehabilitation. Proprioceptive neuromuscular facilitation (PNF) is a therapeutic approach that provides input with cutaneous, proprioceptive, auditory and visual stimuli to provide functional improvement in motor movement and can play a vital role in the rehabilitation of many injuries. PNF is a special manual technique that combines different planes of movement and is applied by physiotherapists to improve the functional status of the patient. This method plays an effective role in supporting the patient to achieve their goals by making movements more functional. Studies have shown that it is effective in pain management, increasing range of motion, developing muscle strength and endurance, improving balance and coordination, providing proximal stability and supporting functional progress. Neuromuscular reeducation applications are widely preferred in the early rehabilitation processes of acute or subacute periods in order to improve motor functions of paralyzed patients. This method stimulates the proprioceptive organs in the muscles and tendons to improve muscle functions, promotes the emergence of postural reflexes, and regulates muscle contraction to increase strength, flexibility, balance, and coordination. Many articles have revealed that a PNF-based program has the potential to produce positive results on motor function in older adults with acute and chronic paralysis. A 2018 study found that PNF was effective in improving upper extremity motor skills and function in stroke patients in the acute and/or subacute stages, while other studies found that it was effective in reducing spasticity, increasing joint range of motion, and improving self-care function in the chronic stage.

Another neuromuscular treatment method used in stroke patients is kinesiology taping. Kinesiology taping (KT) was introduced by Kenzo Kase in 1996 and is a combination of applying appropriate tension along the elastic therapeutic tape and placing the target muscle in a tense position, and is widely used as an interesting and relatively new method for various clinical treatments. KT is a type of elastic, cotton, adhesive bandage with a 140% extensibility that can mimic the elasticity and tension of human skin, muscle, and fascia. Previous studies have shown that kinesiology taping can increase blood circulation, provide mechanical support and proprioceptive feedback, improve joint range of motion, and activate muscles. KT has gained popularity in clinical practice and has been used in clinical practice worldwide. KT applications may promote functional use of the upper and lower extremities by supporting weak muscles, relaxing overstretched muscles, reducing pain and further improving balance ability. Based on these observations, kinesiology taping is considered a potential treatment for spasticity, motor control and tone regulation, providing prorioceptive input and increasing functions. The International Classification of Functioning, Disability and Health (ICF) is an international and standardized classification system developed by the World Health Organization (WHO) to be applied in many branches of health and to evaluate functionality, disability and health holistically. ICF can be used for many purposes, this classification system is a policy and planning tool for decision makers. In addition to being used to categorize health, ICF can be used to determine functional status and to plan rehabilitation programs and guide goal achievement. An interdisciplinary team approach in stroke treatment, where different specialists work together harmoniously and closely, has been described as the basis for effective stroke rehabilitation programs. Measuring, reporting and comparing outcomes across each treatment approach is important to improve outcomes and make informed choices about how to optimize healthcare and rationalize costs.

ELIGIBILITY:
Inclusion Criteria:Inclusion criteria for the study (Junior et al., 2019; Kim & Kim, 2015; Saklecha et al., 2023)

* Stroke diagnosed by MRI or CT, regardless of ischemic or hemorrhagic origin,
* Hemiplegia caused by stroke alone,
* At least 6 and at most 24 months have passed since the stroke was diagnosed
* Being over 18 years of age,
* Volunteering to participate in the study
* Scoring 24 or more on the Standardized Mini Mental State Examination (if illiterate, scoring 18 or more is sufficient)
* Cooperating with evaluation, tests and treatment
* Understanding and speaking Turkish
* Being at least stage 4 according to Brunnstrom staging

Exclusion Criteria:

* Exclusion Criteria (Junior et al., 2019; Kim & Kim, 2015; Saklecha et al., 2023)
* Individuals with bilateral hemiplegia
* Individuals with unstable vital signs
* Individuals with any open wound in the upper extremity
* Pathological conditions affecting upper extremity sensation (undergoing surgery after fracture, etc.)
* Individuals with a BMI value greater than 29.9 kg/m2
* Individuals with a Standardized Mini Mental Test score below 24 points (18 points)
* Individuals with major neurological or rheumatological disorders affecting the musculoskeletal system other than stroke (Polyneuropathy, Parkinson's, Multiple Sclerosis, Rheumatoid Arthritis, etc.)
* Presence of upper extremity amputation
* Being at less than stage 4 according to Brunnstrom staging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
The Fugl Meyer assessment | Beginning of the study and end of week 8 (when 24 sessions are completed)
  The Fugl Meyer assessment scale is a stroke-specific, performance-based scale, and each parameter is scored as 0; unsuccessful, 1; partially successful, and 2; completely successful performance. In the shoulder, elbow, and forearm, reflex activity, voluntary movements performed with dynamic flexor and/or extensor synergies, voluntary movements performed using dynamic flexor and extensor synergies together, voluntary movements performed without or with very little dependence on synergies, and normal reflex activity parameters are evaluated. When evaluating the wrist, three different functions of the wrist muscles are evaluated. In the hemiplegia hand evaluation, 7 movements (flexion, extension, and five grip functions) are evaluated. In the coordination/speed evaluation, a finger-nose test is performed for the upper extremity. During this test, tremor, dysmetria, and speed of movement are evaluated. The maximum motor performance score for the upper extremity is 66 points.
Action Research Arm Test (ARAT) | Beginning of the study and end of week 8 (when 24 sessions are completed)
  The ARAT observes arm and hand movements during the performance of a variety of reaching and grasping tasks. It measures the ability to qualitatively manipulate and carry large or small objects in relation to manual dexterity and proximal strength for the upper extremity. The ARAT rates the upper extremity on a 4-point scale (maximum of 57 points for each upper extremity): 3 points if the task is performed normally; 2 points if the task is completed but takes an abnormally long time; 2 points if performed with great difficulty or poorly coordinated movements; 1 point if the task is only partially completed; and 0 points if the task is not performed at all.
The Box-Block Test | Beginning of the study and end of week 8 (when 24 sessions are completed)
  The Box-Block Test measures unilateral manual dexterity. It is a fast, simple and inexpensive test. It can be used in a wide variety of diseases, including stroke patients. It consists of a box divided into two and 150 blocks. The wooden blocks are cubes measuring 2.5 cm x 2.5 cm x 2.5 cm. The barrier in the middle of the box is 15.2 cm. Patients are asked to throw the blocks from one section to the other, one by one, within 60 seconds and the number of blocks is recorded.
Nine hole Peg Test | Beginning of the study and end of week 8 (when 24 sessions are completed)
  It is a simple and quick test used to evaluate changes in hand functions. The participant is asked to insert nine rods into a wooden block with nine holes as quickly as possible and then remove them. The test is repeated twice and the score is determined as the average of the two trials. The participant is expected to perform the test with the hand on the affected side of the body.

SECONDARY OUTCOMES:
Environmental Quality Scale | Beginning of the study and end of week 8 (when 24 sessions are completed)
  The scale evaluates the impact of the environment on the individual's abilities and limitations while performing daily activities. The short form consists of 26 questions in total. Each question includes two options: facilitating and challenging.
  The scale's scoring ranges from -3 to 3. The facilitating option includes a score of 1 to 3, and the challenging option includes a score of -1 to -3. A score between 1 and 3 indicates that environmental factors facilitate the individual's daily life and social roles, and a score of zero indicates that they have no effect on social interaction. A score between -1 and -3 is considered negative. All positive and negative results are added up separately. The application takes approximately 10 minutes.
Upper Extremity Motor Activity Diary-28 | Beginning of the study and end of week 8 (when 24 sessions are completed)
  This scale, which aims to evaluate the function of the hemiparetic upper extremity, was developed by Uswatte et al. in 2006. 30 upper extremity functions are evaluated and scored with 2 different scales as "level of use" and "quality of use". The scores for each scale are calculated by adding them up and dividing them by the number of marked items. The validity and reliability of the scale in Turkish has been done.
Social Adaptation Scale | Beginning of the study and end of week 8 (when 24 sessions are completed)
  The social adaptation scale is a scale consisting of 10 items (34). The survey focuses on personal experiences, perspectives and personal satisfaction with the level of integration with society rather than the objective and observable aspects of social integration.

CONTACTS AND LOCATIONS:
Overall Officials: Berrak Varhan, Study Director — Istinye University; Mahmut Yaran, Study Director — Ondokuz Mayıs University
Locations (2):
- Turkey (Türkiye) (2):
  - İstinye University, Bahçeşehir Liv Hospital, Istanbul, Bahçeşir
  - Ondokuz Mayıs Üniversitesi, SUVAM Havza Fizik Tedavi ve Rehabilitasyon Merkezin, Samsun, Havza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] EFFECTIVENESS OF THE PROPRIOCEPTIVE NEUROMUSCULAR FACILITATION METHOD APPLICATION ON UPPER LIMB FUNCTIONS IN PATIENTS AFTER STROKE: A SYSTEMATIC REVIEW OF LITERATURE
- See also: Effectiveness of the proprioceptive neuromuscular facilitation method application on upper lımb functions in patients after stroke: a systematic review of literature — https://journals.rta.lv/index.php/SIE/article/view/7793
- See also: Factors associated with post-stroke social participation: A quantitative study based on the ICF framework — https://pubmed.ncbi.nlm.nih.gov/35779831/
- See also: Effectiveness of kinesio taping for chronic stroke patients: a systematic review with meta-analysis — https://pubmed.ncbi.nlm.nih.gov/37530391/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-01-01): https://cdn.clinicaltrials.gov/large-docs/96/NCT07014696/Prot_SAP_000.pdf
  • Informed Consent Form (2025-01-01): https://cdn.clinicaltrials.gov/large-docs/96/NCT07014696/ICF_001.pdf